CLINICAL TRIAL: NCT03798977
Title: Preclinical Validation of New Anti-melanoma Compounds: Study on Patient Melanoma Cells Sensitive and Resistant to BRAF/MEK Inhibitors
Brief Title: Preclinical Validation of New Anti-melanoma Compounds
Acronym: ERMELATHER
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Nice (Other)
Responsible Party: Sponsor
Other Study IDs: 17-PRTK-01
Record Dates: First submitted 2018-12-27; First posted 2019-01-10 (Actual); Last update posted 2024-02-06 (Actual); Status verified 2024-02

CONDITIONS: Melanoma
Keywords: Skin metastasis; Resistance; Endoplasmic reticulum stress; Metastasis
MeSH Terms: conditions — Melanoma; Neoplasm Metastasis

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — biopsy of a target lesion (skin, lymph node or visceral metastases)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This research program is in keeping with the chemistry/biology/clinical interface and gathers 4 teams with complementary expertise in these respective fields. It will allow deciphering the mechanism(s) of action of new Thiazole-Benzenesulfonamide family (TZB) derivatives on metastatic melanoma sensitive and resistant to BRAF and MEK inhibitors. Investigators will use melanoma cell lines and primary cells from patients to validate these compounds in collaboration with clinical team 2 and 4. In conclusion, the investigators expect to establish the proof of concept that this new class of bioactive molecules (first in class) we developed in collaboration with Team 3 have the potential to go to the clinic for the treatment of highly aggressive cancers and particularly metastatic melanoma sensitive and resistant B-Raf and MEK inhibitors. Furthermore, the realization of this project can undoubtedly increase the knowledge of mechanisms and signaling pathways that are involved in resistant to BRAF and MEK inhibitors, and allow the selection of drug candidates capable of restoring the sensitivity of these melanoma cells.

ELIGIBILITY:
Inclusion Criteria:

* Patient with metastatic melanoma
* Not opposition of the patient will have been looked for

Exclusion Criteria:

* Primary resistance,
* Absence of resistance,
* Patient already included in other trials

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient with metastatic melanoma
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2018-02-01 (Actual); Primary Completion 2021-07-31 (Actual); Study Completion 2021-07-31 (Actual)

PRIMARY OUTCOMES:
BRAF mutation | 24 months
  The status of the BRAF mutation will be expressed through laboratory analysis of the samples collected, i.e. positive or negative.

CONTACTS AND LOCATIONS:
Locations (1):
- Nice hospital, Nice, France

IPD SHARING:
Plan to Share IPD: Undecided